CLINICAL TRIAL: NCT03668730
Title: A Phase II Trial of Induction Chemotherapy Followed by Cisplatin With Low Dose vs. Standard Dose IMRT in Stage III Nasopharyngeal Carcinoma Patients With Pretreatment EBV DNA<4000 Copy/ml
Brief Title: Reduced-dose Radiotherapy for Low-risk Stage III Patients With Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-020-01
Record Dates: First submitted 2018-06-08; First posted 2018-09-13 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; IMRT; Radiation dose; induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced dose group (Experimental): After 2 cycles of induction chemotherapy with Paclitaxel Liposome, Cisplatin and 5-Fluorouracil, patients undergo low-dose intensity-modulated radiotherapy (IMRT) 5 days per week for approximately 6 weeks (30 fractions). Patients also receive cisplatin once per three week for 3 cycles.
  Interventions: Radiation: Intensity-modulated radiation therapy; Drug: Paclitaxel liposome; Drug: Cisplatin; Drug: 5-Fluorouracil
- Standard dose group (Experimental): After 2 cycles of induction chemotherapy with Paclitaxel Liposome,Cisplatin and 5-Fluorouracil, patients undergo standard-dose intensity-modulated radiotherapy (IMRT) 5 days per week for approximately 6 weeks (33 fractions). Patients also receive cisplatin once per three week for 3 cycles.
  Interventions: Radiation: Intensity-modulated radiation therapy; Drug: Paclitaxel liposome; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy — Patients undergo low-dose OR standard dose IMRT based on their radiographic response to induction chemotherapy
Drug: Paclitaxel liposome — Patients receive Paclitaxel liposome by 135mg/m2 with a total of two cycles.
Drug: Cisplatin — Patients receive Cisplatin by 25mg/m2 on day1-day3 with a total of two cycles as induction chemotherapy ; patients receive cisplatin by 100mg/m2 with a total of three cycles as concurrent chemotherapy.
Drug: 5-Fluorouracil — Patients receive 5-Fluorouracil by 3750mg/m2 civ120h with a total of three cycles.

SUMMARY:
To study the 2-year PFS (progression-free survival) of patients with stage III nasopharyngeal carcinoma of pretreatment EBV DNA<4000 copy/ml treated with induction chemotherapy followed by two different doses of intensity-modulated radiation therapy and cisplatin.

DETAILED DESCRIPTION:
To explore the 2 year PFS of patients with stage III nasopharyngeal carcinoma of pretreatment EBV DNA<4000 copy/ml treated with induction chemotherapy followed by reduced-dose radiation and cisplatin. The enrolled patients will receive 2 cycles of TPF regimen induction chemotherapy, if radiographic CR/PR and EBV DNA=0 after induction chemotherapy, the patients will be delivered by 60 Gy IMRT combined with 3 cycles of cisplatin concurrent chemotherapy. If radiographic SD/PD or EBV DNA>0 after induction chemotherapy, the patients will receive a total of 70 Gy IMRT combined with 3 cycles of cisplatin concurrent chemotherapy.

The included patients will be treated with 2 cycles of TPF regimen induction chemotherapy and 60Gy IMRT combined with cisplatin concurrent chemotherapy. The TPF regimen is consist of paclitaxel liposome 135mg/m2 d1, cisplatin 25mg/m2d1-d3 and 5-Fu 3750mg/m2 civ120h, with a total of two cycles. Concurrent cisplatin chemotherapy is delivered with dose of 100mg/m2, a total of three cycles. The third cycle of cisplatin concurrent chemotherapy is allowed to be delivered within one week after IMRT finished.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of NPC(WHO II or III).
2. Stage III（8thAJCC/UICC staging system) and pretreatment EBVDNA<4000opies/ml.
3. Aged 18-70 years。
4. ECOG = 0-1。
5. HGB≥90 g/L，WBC≥4×109 /L，PLT≥100×109 /L.
6. ALT,AST<2.5 fold of ULN；TBIL<2.0×ULN。
7. CCR≥60ml/min or Cr<1.5×ULN。
8. Signed informed consent

Exclusion Criteria:

1. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
2. Age <18 or >70years.
3. Treatment with palliative intent.
4. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
5. Pregnancy or lactation.
6. History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
7. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
8. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS(progression free survival) | 2 years
  Defined from date of registration to date of first documentation of progression and/or distant metastasis,or death due to any cause. The primary study population for this endpoint is patients who were confirmed post-induction CR /PR and EBV DNA=0 and subsequently received 60Gy radiation therapy.

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 years
  Defined from date of registration to date of first documentation of death from any cause or censored at the date of the last follow-up.
Locoregional relapse-free survival(LRFS) | 2 years
  Defined from date of registration to date of first documentation of locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 2 years
  Defined from date of registration to date of first documentation of distant metastases or until the date of the last follow-up visit.
Overall response rate | 2 years
  Tumour response rate was classified according to RECIST, version 1.1
Incidence of acute toxicity | 2 years
  Numbers of patients of treatment-related adverse events as assessed by CTCAE v4.0.
Incidence of late toxicity | 2 years
  Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Change of ADC( apparent diffusion coefficient ) value of DWI(Diffusion-Weighted MRI) of patients predictive of failure | 2 years
  The ADC value of each patient of Diffusion-Weighted MRI at pretreatment and after induction chemotherapy was calculated were evaluated independently on a work station.
Change of QoL | 1 years
  QoL scores were assessed for each scale by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) before induction chemotherapy, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy.
Change of EORTC quality of life questionnaire(QLQ) Head and Neck score | 1 years
  QoL scores were assessed by using EORTC quality of life questionnaire(QLQ) Head and Neck. The QLQ-H&N35 is composed of seven multi-item symptom scales (pain, swallowing, sensation, speech, eating from a social,perspective, social interactions, and sexuality) and 11 single-item symptom scales (teeth, opening mouth,dry mouth, sticky saliva, coughing, felt ill, pain medication use, nutritional supplementation, feeding tube requirement, weight loss, and weight gain). All of the scales and items ranged in score from 0 to 100. A high score for a functional or global QoL scale represents a relatively high/healthy level of functional or global QoL, whereas a high score for a symptom scale or item represents a high number of symptoms or problems.
Plasma EBV DNA copy number | 2 years
  Plasma EBV DNA copy number with either reduced or standard dose radiotherapy was assessed by qRT-PCR at pretreatment. The predictive value of plasma EBV DNA copy number was assessed by survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Qiang Mai, MD.PHD, Study Chair — Sun Yat-sen University
Locations (1):
- Hai Qiang Mai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo SS, Yang JH, Sun XS, Liu LZ, Yang ZC, Liu LT, Liu SL, Li XY, Lv XF, Luo DH, Li JB, Liu Q, Wang P, Guo L, Mo HY, Sun R, Yang Q, Liang YJ, Jia GD, Zhao C, Chen QY, Tang LQ, Mai HQ. Reduced-dose radiotherapy for Epstein-Barr virus DNA selected staged III nasopharyngeal carcinoma: A single-arm, phase 2 trial. Eur J Cancer. 2023 Nov;194:113336. doi: 10.1016/j.ejca.2023.113336. Epub 2023 Sep 9. PMID 37801967